CLINICAL TRIAL: NCT00297167
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Treatment, Crossover Study to Evaluate the Safety and Efficacy of Eurand Pancreatic Enzyme Product (PEP) in Patients With Cystic Fibrosis and Exocrine Pancreatic Insufficiency
Brief Title: Study to Evaluate the Safety and Efficacy of EUR-1008 (APT-1008) Pancreatic Enzyme Product in Participants With Cystic Fibrosis and Exocrine Pancreatic Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EUR-1008-M
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: CF; Cystic Fibrosis; EPI; Exocrine Pancreatic Insufficiency; Pancreatic; Enzyme; PEP
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

ARMS (2):
- EUR-1008 (APT-1008) First, Then Placebo (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008); Drug: Placebo
- Placebo First, Then EUR-1008 (APT-1008) (Experimental)
  Interventions: Drug: Placebo; Drug: EUR-1008 (APT-1008)

INTERVENTIONS:
Drug: EUR-1008 (APT-1008) — EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule will be given orally daily in first double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). The capsules could be opened and sprinkled on acidic food and half of the established dose was used with snacks. Treatment duration for first double-blind intervention period will be 2 days home treatment and 3 to 5 days hospital treatment.
  Arms: EUR-1008 (APT-1008) First, Then Placebo
Drug: Placebo — Placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule will be given orally daily in second double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). Treatment duration for second double-blind intervention period will be 2 days home treatment and 3 to 5 days hospital treatment.
  Arms: EUR-1008 (APT-1008) First, Then Placebo
Drug: Placebo — Placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule will be given orally daily in first double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). Treatment duration for first double-blind intervention period will be 2 days home treatment and 3 to 5 days hospital treatment.
  Arms: Placebo First, Then EUR-1008 (APT-1008)
Drug: EUR-1008 (APT-1008) — EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule will be given orally daily in second double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). Treatment duration for second double-blind intervention period will be 2 days home treatment and 3 to 5 days hospital treatment.
  Arms: Placebo First, Then EUR-1008 (APT-1008)

SUMMARY:
The primary efficacy objective of this study is to compare the coefficient of fat absorption (CFA) following oral administration of Aptalis Pharma's (formerly Eurand Pharmaceuticals) pancreatic enzyme product (PEP) capsules and placebo in participants with cystic fibrosis (CF) and exocrine pancreatic insufficiency (EPI).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 2-treatment, crossover, multicenter trial in participants with CF and EPI. The study consists of a screening period (1 to 14 days), a washout period (2 days), a dose titration/stabilization period (6 to 9 days), a blinded randomized treatment period (6 to 7 days), an open-label normalization period 1 (5 to 14 days), a blinded crossover treatment period (6 to 7 days), followed by an open-label normalization period 2 (7 days). The order of treatments (placebo followed by EUR-1008 [APT-1008] or EUR-1008 [APT-1008] followed by placebo) will be determined by randomization at the beginning of randomization treatment period only and will be carried through the crossover treatment period. The starting dose will be 1,000 lipase units per kilogram per meal (lipase units/kg/meal), which will be titrated to control symptoms of EPI, with the total dose not exceeding 10,000 lipase units/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age greater than or equal to (>=) 7 years at the time of enrollment
* Participants with weight 70 kg or less and be in an adequate nutritional status as indicated by a body mass index (BMI) >=20 kg/m^2 for ages 18 and above, or a BMI above the twenty fifth percentile for participants aged 7 to 17 years
* Participants with confirmed diagnosis of CF who have 2 clinical features consistent with CF, and have either a genotype with 2 identifiable mutations consistent with CF or a sweat chloride concentration that is more than 60 milliequivalent per liter by quantitative pilocarpine iontophoresis
* Participants with confirmed diagnosis of EPI who are currently receiving treatment with a commercially available PEP and have documented with a fecal elastase of <100 microgram per gram stool (if no documentation was available, a stool sample was taken at Screening for determination of fecal elastase).
* Clinically stable participants with no evidence of acute respiratory disease or any other acute condition
* Participants who are willing and able to interrupt current CF treatment for CF-related malabsorption along with any medications that may affect gastric motility or stomach power of hydrogen (pH)
* Participants 18 years of age and older had to a) understand the requirements of the study, b) provide written informed consent, c) agree to abide by the study restrictions, and d) return for the required assessments
* Participants 7 to 17 years of age must have a parent(s) or legal guardian who provides written informed consent, agree to abide by the study restrictions
* Females participants of childbearing potential must have a negative serum pregnancy test at screening and must agree to use adequate birth control during the study

Exclusion Criteria:

* Participants with fibrosing colonopathy, hyperuricemia or hyperuricosuria
* Participants who are allergic to pork or other porcine PEPs
* Participants with forced expiratory volume (FEV1) <30 percent of predicted FEV1 at screening
* Participants with any acute systemic administration of an antibiotic for any reason in the previous 4 weeks; however, a low stable dose of an antibiotic or chronic treatment with an inhalatory antibiotic is allowed
* Participants with hepatic insufficiency as defined by history or presence of ascites or serum albumin level of < 3.0 milligram/deciliter, or a coagulopathy with an international normalized ratio that is greater than 1.7
* Participants who have used an acute dose of any steroid in the previous 2 weeks; however, low chronic doses of a steroid is allowed
* Participants with history of or current diagnosis of distal ileal obstruction syndrome (DIOS) as evidenced or suggested by constipation, abdominal pain, anorexia, early satiety, recurrent vomiting, and palpable fecal mass on physical examination (the absence of DIOS will be confirmed by an X-ray of the abdomen taken at screening)
* Participants with any solid organ transplant or surgery affecting the bowel. Participants with a history of appendectomy and inguinal (non-incarcerated) hernioplasty or meconium ileus without the need for bowel resection could be enrolled. Gastrointestinal-tube-fed patients, in absence of dumping syndrome, were also eligible
* Participants with history of or current screening evaluation of hyperglycemia as defined by an 8-hour fasting blood glucose (FBG) of >126 mg/dL, or of CF-related diabetes as determined according to the Cystic Fibrosis Foundation (CFF) Consensus Conference of January 1999 (Section IX Part II), that is: a) FBG >126 mg/dL (7.0 millimoles per liter [mmol/L]) on two or more occasions b)FBG >126 mg/dL (7.0 mmol/L) plus casual (without regard to time of day or last meal consumed) glucose level >200 mg/dL (11.1 mmol/L) c)Casual (previously called random) glucose levels >200 mg/dL (11.1 mmol/L) on two or more occasions with symptoms
* Participants using an enzyme preparation in excess of 10,000-lipase units/kg/day
* Participants using an immunosuppressive drug
* Participants who are expecting an inability to tolerate the washout period and/or the placebo treatment
* Participants participating in an investigational study of a drug, biologic, or device not currently approved for marketing, within 30 days of screening visit
* Female participants who are pregnant or breastfeeding, or unwilling to use effective birth control during study
* Participants with any condition that would, in the investigator's opinion, limit the participant's ability to complete the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (1):
- University of Texas Health Center at Tyler, Tyler, Texas, United States

REFERENCES:
- [Derived] Wooldridge JL, Heubi JE, Amaro-Galvez R, Boas SR, Blake KV, Nasr SZ, Chatfield B, McColley SA, Woo MS, Hardy KA, Kravitz RM, Straforini C, Anelli M, Lee C. EUR-1008 pancreatic enzyme replacement is safe and effective in patients with cystic fibrosis and pancreatic insufficiency. J Cyst Fibros. 2009 Dec;8(6):405-17. doi: 10.1016/j.jcf.2009.07.006. Epub 2009 Aug 15. PMID 19683970

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 34 participants who were enrolled and treated during open-label dose titration and stabilization period, 1 participant withdrew from the study before randomization to first double-blind intervention period.
Groups:
- Placebo First, Then EUR-1008 (APT-1008): Placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule and was given orally daily in the first double-blind intervention period followed by EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule and was given orally daily in the second double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). The capsules could be opened and sprinkled on acidic food and half of the established dose was used with snacks. Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment. The stabilized dose was not to exceed 10,000 lipase units per kilogram body weight per day (lipase units/kg/day).
- EUR-1008 (APT-1008) First, Then Placebo: EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule and was given orally daily in the first double-blind intervention period followed by placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule and was given orally daily in the second double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). The capsules could be opened and sprinkled on acidic food and half of the established dose was used with snacks. Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment. The stabilized dose was not to exceed 10,000 lipase units/kg/day.
- EUR-1008 (APT-1008) (Open-label): EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule and was given orally daily at a fixed stabilized dose during open-label normalization period 1 (5 to 14 days) after first double-blind interventional period and during open-label normalization period 2 (7 days) after second double-blind interventional period.
Period: First Double-blind Intervention Period
Arm/Group | Placebo First, Then EUR-1008 (APT-1008) | EUR-1008 (APT-1008) First, Then Placebo | EUR-1008 (APT-1008) (Open-label)
Started | 17 | 16 | 0
Completed | 17 | 16 | 0
Not Completed | 0 | 0 | 0
Period: Open-label Dose Normalization Period 1
Arm/Group | Placebo First, Then EUR-1008 (APT-1008) | EUR-1008 (APT-1008) First, Then Placebo | EUR-1008 (APT-1008) (Open-label)
Started | 0 | 0 | 33
Completed | 0 | 0 | 32
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Second Double-blind Intervention Period
Arm/Group | Placebo First, Then EUR-1008 (APT-1008) | EUR-1008 (APT-1008) First, Then Placebo | EUR-1008 (APT-1008) (Open-label)
Started | 17 | 15 | 0
Completed | 16 | 15 | 0
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Open-label Dose Normalization Period 2
Arm/Group | Placebo First, Then EUR-1008 (APT-1008) | EUR-1008 (APT-1008) First, Then Placebo | EUR-1008 (APT-1008) (Open-label)
Started | 0 | 0 | 31
Completed | 0 | 0 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study treatment.
Groups:
- Entire Study Population: Includes participants who received EUR-1008 (APT-1008) in open-label dose titration and stabilization phase; and EUR-1008 (APT-1008) first and placebo first after randomization to study treatment.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Coefficient of Fat Absorption (CFA%)
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)multiplied by 100, determined in the stools collected during the 72-hour hospitalization period. Mean percent CFA was calculated for Day 3 to Day 6 during hospital treatment in first and second double-blind (DB) intervention periods.
Time Frame: Day 3 up to Day 6 of hospital treatment in first and second double-blind intervention periods
Population: Efficacy analysis population included all randomized and treated participants with at least 1 post-baseline measurement for each double-blind intervention period. Here "N" (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent CFA
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule and was given orally daily in the first and second double-blind intervention periods; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). The capsules could be opened and sprinkled on acidic food and half of the established dose was used with snacks. Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment. The stabilized dose was not to exceed 10,000 lipase units/kg/day.
- Placebo: Placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule and was given orally daily in the first and second double-blind intervention periods; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment.
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 31
percent CFA | 88.28 (2.599) | 62.76 (2.639)
Statistical Analysis 1: Comparison: EUR-1008 (APT-1008) vs Placebo; P-Value was calculated using analysis of variance (ANOVA) model which included main effects for treatment and sequence and participant nested in sequence as a random effect; Test type: Superiority or Other; p < 0.001, ANOVA; Least Square (LS) Mean Difference = -25.52, 95% CI 2-sided [-31.73 to -19.32]

2. Secondary Outcome: Percent Coefficient of Nitrogen Absorption (CNA%)
Description: Percent CNA was calculated as ([nitrogen intake-nitrogen excretion]/nitrogen intake)*100, determined in the stools collected during the 72-hour hospitalization period. Nitrogen intake was calculated as protein intake/6.2. Nitrogen excretion was measured as total fecal nitrogen. Mean percent CNA was calculated for Day 3 to Day 6 during hospital treatment in first and second double-blind intervention periods.
Time Frame: Day 3 up to Day 6 of hospital treatment in first and second double-blind intervention periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent CNA
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 31
percent CNA | 87.17 (2.179) | 65.67 (2.213)
Statistical Analysis 1: Comparison: EUR-1008 (APT-1008) vs Placebo; P-Value was calculated using analysis of variance (ANOVA)model which included main effects for treatment and sequence and participant nested in sequence as a random effect; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = -21.50, 95% CI 2-sided [-26.85 to -16.14]

3. Secondary Outcome: Lipid Levels
Description: Lipid levels were reported for total cholesterol (TC) and high-density lipoprotein cholesterol (HDL-C) from fasted blood and urine samples. Mean lipid levels for Day 6 during first and second double-blind intervention periods were calculated.
Time Frame: End of treatment (Day 6 during first and second double-blind intervention periods)
Population: Safety population included all participants who received at least 1 dose of study treatment. Here "N" (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at specific time point in each treatment arm.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 33 | 30
milligram/deciliter (mg/dL)
  TC: End of Treatment (n=33, 30) | 128.8 (28.98) | 109.1 (29.76)
  HDL-C: End of Treatment (n=33, 30) | 45.5 (10.85) | 37.2 (9.23)

4. Secondary Outcome: Vitamin A Levels
Description: Mean Vitamin A levels for Day 6 during first and second double-blind intervention periods were calculated.
Time Frame: End of treatment (Day 6 during first and second double-blind intervention periods)
Population: Safety population included all participants who received at least 1 dose of study treatment. Here "N" (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 33 | 30
microgram per liter (mcg/L) | 422.3 (111.67) | 363.2 (100.33)

5. Secondary Outcome: Vitamin E Levels
Description: Mean Vitamin E levels for Day 6 during first and second double-blind intervention periods were calculated.
Time Frame: End of treatment (Day 6 during first and second double-blind intervention periods)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 33 | 30
mg/L | 8.25 (3.115) | 6.69 (2.648)

6. Secondary Outcome: Mean Daily Number of Stools
Description: Mean daily number of stools of each participant was calculated from frequency of stools by the participant per day. Mean daily number of stools during the collection period (Day 3 to Day 6 in first and second double-blind intervention periods) for total participants was summarized.
Time Frame: Day 3 up to Day 6 during first and second double-blind intervention periods
Population: Efficacy analysis population included all randomized and treated participants with at least 1 post-baseline measurement for each double-blind intervention period.
Measure: Mean (Standard Deviation); unit: stools per day
Groups:
- Placebo: Placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule and was given orally daily in the first and second intervention periods; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment.
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 32
stools per day | 1.76 (0.898) | 2.66 (1.418)

7. Secondary Outcome: Percentage of Stool Categorized as Per Consistency
Description: Stool consistency was categorized as hard, formed/normal, soft, watery, or overt diarrhea. Percentage of stools of a specific consistency for each participant at first and second double-blind intervention periods was calculated. Mean percentage of stool consistency during the collection period (Day 3 to Day 6 in first and second intervention periods) for total participants was summarized.
Time Frame: Day 3 up to Day 6 during first and second double-blind intervention periods
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 32
percentage of stools
  Hard | 16.54 (29.637) | 6.24 (18.845)
  Formed/Normal | 53.86 (37.253) | 33.25 (34.414)
  Soft | 29.24 (34.096) | 57.11 (36.105)
  Watery | 0.36 (1.421) | 2.59 (4.836)
  Overt diarrhea | 0.00 (0.000) | 0.82 (3.670)

8. Secondary Outcome: Mean Number of Abdominal Symptoms
Description: Abdominal symptoms included abdominal pain, flatulence and bloating. Symptoms were classified by severity as mild (no impairment of daily activities), moderate (slight impairment of daily activities), or severe (unable to perform daily activities). Mean number of symptom of specific severity per day for each participant was calculated. Mean number of symptoms per day was calculated for Day 3 to Day 6 in first and second double-blind intervention periods for total participants.
Time Frame: Day 3 up to Day 6 during first and second double-blind intervention periods
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: symptoms per day
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 32
symptoms per day
  Bloating: Mild | 0.10 (0.300) | 0.31 (0.718)
  Bloating: Moderate | 0.05 (0.191) | 0.10 (0.329)
  Bloating: Severe | 0.00 (0.000) | 0.09 (0.495)
  Flatulence: Mild | 0.40 (0.688) | 0.70 (1.134)
  Flatulence: Moderate | 0.08 (0.275) | 0.41 (1.160)
  Flatulence: Severe | 0.00 (0.000) | 0.18 (0.719)
  Pain: Mild | 0.16 (0.433) | 0.62 (0.901)
  Pain: Moderate | 0.08 (0.379) | 0.32 (0.754)
  Pain: Severe | 0.00 (0.022) | 0.09 (0.228)

9. Other Pre Specified Outcome: Percentage of Visible Oil or Grease in Stool
Description: Mean percentage of stools with visible oil or grease during the collection period (Day 3 to Day 6 in first and second intervention periods) for total participants was summarized. Percentage was calculated as the number of stools with visible oil or grease divided by the total number of stool per day.
Time Frame: Day 3 up to Day 6 of hospital treatment in first and second double-blind intervention periods
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of visible oil or grease/day
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 32
percentage of visible oil or grease/day | 6.78 (17.354) | 27.97 (33.571)

10. Other Pre Specified Outcome: Percentage of Stools With Blood
Description: Mean percentage of stools with blood during the collection period (Day 3 to Day 6 in first and second intervention periods) for total participants was summarized. Percentage was calculated as the number of stools with blood divided by the total number of stool per day.
Time Frame: Day 3 up to Day 6 of hospital treatment in first and second double-blind intervention periods
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of stools with blood per day
Arm/Group | EUR-1008 (APT-1008) | Placebo
Number analyzed (Participants) | 32 | 32
percentage of stools with blood per day | 0.17 (0.174) | 1.13 (4.647)

ADVERSE EVENTS:
Description: Adverse event (AE) was defined as any untoward medical occurrence regardless of causal relationship to study medication. Serious adverse event (SAE) was any event that resulted in death,life threatening,required or prolonged in-patient hospitalization,significant disability/incapacity,or was a congenital anomaly/birth defect or assessed as important medical event.
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) microtablets (5000 lipase units) or minitablets (10000, 15000 or 20000 lipase units) contained in a capsule was given orally daily in the first and second double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). The capsules could be sprinkled on acidic food and half of the established dose was used with snacks. Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment. Participants received EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule was given orally daily at a fixed stabilized dose for 5 to 14 days during open-label dose normalization period 1 and for 7 days during open-label dose normalization period 2 which was maintained after each double-blind intervention period. The stabilized dose was not to exceed 10,000 lipase units per kilogram body weight per day (units/kg/day).
- Placebo: Placebo matched to EUR-1008 (APT-1008) microtablets or minitablets contained in a capsule was given orally daily in the first and second double-blind intervention period; at a dose based on investigator's discretion as achieved during dose titration and stabilization period (6 to 9 days). Treatment duration for each double-blind intervention period was 2 days home treatment and 3 to 5 days hospital treatment.
Arm/Group | EUR-1008 (APT-1008) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/34 | 0/32
Other Adverse Events (participants affected / at risk) | 19/34 | 16/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EUR-1008 (APT-1008) (N=34) | Placebo (N=32)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — SAEs for EUR-1008 occurred during the first open-label dose stabilization period, during which all participants were on EUR-1008.
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — SAEs for EUR-1008 occurred during the first open-label dose stabilization period, during which all participants were on EUR-1008.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EUR-1008 (APT-1008) (N=34) | Placebo (N=32)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Abdominal distension (Gastrointestinal disorders) | 2 | 3 — These data represent AEs collected during both double blind treatment periods.
Abdominal pain (Gastrointestinal disorders) | 4 | 6 — These data represent AEs collected during both double blind treatment periods.
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 — These data represent AEs collected during both double blind treatment periods.
Abnormal faeces (Gastrointestinal disorders) | 1 | 3 — These data represent AEs collected during both double blind treatment periods.
Flatulence (Gastrointestinal disorders) | 2 | 3 — These data represent AEs collected during both double blind treatment periods.
Frequent bowel movements (Gastrointestinal disorders) | 1 | 2 — These data represent AEs collected during both double blind treatment periods.
Nausea (Gastrointestinal disorders) | 1 | 1 — These data represent AEs collected during both double blind treatment periods.
Steatorrhoea (Gastrointestinal disorders) | 0 | 4 — These data represent AEs collected during both double blind treatment periods.
Vomiting (Gastrointestinal disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Early satiety (General disorders) | 2 | 0 — These data represent AEs collected during both double blind treatment periods.
Contusion (Injury, poisoning and procedural complications) | 2 | 0 — These data represent AEs collected during both double blind treatment periods.
Injury (Injury, poisoning and procedural complications) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Weight decreased (Investigations) | 2 | 2 — These data represent AEs collected during both double blind treatment periods.
Headache (Nervous system disorders) | 5 | 0 — These data represent AEs collected during both double blind treatment periods.
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — These data represent AEs collected during both double blind treatment periods.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Bowel sounds abnormal (Gastrointestinal disorders) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Constipation (Gastrointestinal disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Chest pain (General disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Oedema mucosal (General disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Pyrexia (General disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Otitis externa (Infections and infestations) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Anal injury (Injury, poisoning and procedural complications) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Fall (Injury, poisoning and procedural complications) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Anorexia (Metabolism and nutrition disorders) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Dizziness (Nervous system disorders) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Vaginal burning sensation (Reproductive system and breast disorders) | 0 | 1 — These data represent AEs collected during both double blind treatment periods.
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — These data represent AEs collected during both double blind treatment periods.
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.
Haematoma (Vascular disorders) | 1 | 0 — These data represent AEs collected during both double blind treatment periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions may vary in accordance with each agreement that is negotiated with individual investigators. Sponsor will allow publication after multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and defer publication for period of time to allow Sponsor to obtain patent or other intellectual property right protection.